CLINICAL TRIAL: NCT03977337
Title: Perioperative Pulmonary Monitoring in Major Emergency Surgery -the PROMIES Project
Brief Title: Perioperative Pulmonary Monitoring in Major Emergency Surgery
Acronym: PROMIES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PROMIES
Record Dates: First submitted 2019-01-14; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Pulmonary Complication; Cardiovascular Complication; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Major emergency abdominal surgery — Major emergency gastrointestinal surgery performed within 72 hours of an acute admission or an acute reoperation.

SUMMARY:
1. Describe the incidence of postoperative hypoxemia after major emergency abdominal surgery as well as correlate this to clinical outcomes.
2. Investigate the association between postoperative pulmonary complications and respiratory muscle dysfunction.
3. Investigate the association between the length and type of incision as well as the distance to the xiphoid process and respiratory muscle dysfunction.
4. Investigate the association between postoperative hypoxemia, myocardial ischemia and ischemic electrocardiographic (ECG) changes within three days of major emergency abdominal surgery
5. Describe the incidence of postoperative cardiac arrhythmias within three days of major emergency abdominal surgery and the association with postoperative cardiovascular complications within 30 days, 90 days and 1 year of surgery.
6. Describe the association between HRV and postoperative cardiovascular and non-cardiovascular complications within 30 days, 90 days and 1 year of surgery

ELIGIBILITY:
Inclusion Criteria:

* Surgery within 72 hours of an acute admission to the Department of Surgery or an acute reoperation.
* Major gastrointestinal surgery on the gastrointestinal tract.

This will include:

* Open, laparoscopic, or laparoscopically-assisted procedures
* Procedures involving the stomach, small or large bowel, or rectum for conditions such as perforation, ischemia, abdominal abscess, bleeding or obstruction
* Washout/evacuation of intra-peritoneal abscess (unless due to appendicitis or cholecystitis - excluded, see below)
* Washout/evacuation of intra-peritoneal hematoma
* Bowel resection/repair due to incarcerated umbilical, inguinal and femoral hernias (but not hernia repair without bowel resection/repair)
* Bowel resection/repair due to obstructing/incarcerated incisional hernias provided the presentation and findings were acute
* Laparotomy/laparoscopy with inoperable pathology (e.g. peritoneal/hepatic metastases)
* Laparoscopic/Open adhesiolysis
* Return to theatre for repair of fascial dehiscence
* Any reoperation/return to theatre meeting the criteria above is included

If multiple procedures (primary surgery or reoperation) are performed on different anatomical sites within the abdominal/pelvic cavity, the patient would be included if the major procedure is general surgical.

Exclusion Criteria:

* Not capable of giving informed consent after oral and written information
* Previously included in the trial
* Elective laparoscopy
* Diagnostic laparotomy/laparoscopy where no subsequent procedure is performed (NB, if no procedure is performed because of inoperable pathology, then include)
* Appendectomy +/- drainage of localized collection unless the procedure is incidental to a non-elective procedure on the GI tract
* Cholecystectomy +/- drainage of localized collection unless the procedure is incidental to a non-elective procedure on the GI tract (All surgery involving the appendix or gallbladder, including any surgery relating to complications such as abscess or bile leak is excluded)
* Non-elective hernia repair without bowel resection.
* Minor abdominal wound dehiscence unless this causes bowel complications requiring resection
* Ruptured ectopic pregnancy, or pelvic abscesses due to pelvic inflammatory disease
* Laparotomy/laparoscopy for pathology caused by blunt or penetrating trauma
* Laparotomy/laparoscopy for esophageal pathology
* Laparotomy/laparoscopy for pathology of the spleen, renal tract, kidneys, liver, gall bladder and biliary tree, pancreas or urinary tract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the department of Surgery, Zealand University Hospital, Denmark.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in postoperative maximal inspiratory mouth pressure from POD1 to POD3 | 3 days
  Maximal inspiratory mouth pressure [cmH2O] is measured on the first and third postoperative day to asses the change
Change in postoperative maximal expiratory mouth pressure from POD1 to POD3 | 3 days
  Maximal expiratory mouth pressure [cmH2O] is measured on the first and third postoperative day to asses the change
Length of surgical incision | Day 1
  The length of the surgical incision [cm] will be measured on the first postoperative day
Heart Rate Variability (HRV) | 3 days
  HRV assessed preoperatively - POD3, if this is not achievable then from POD0 - POD3
The occurence of per- and postoperative cardiac arrhythmias (until POD3) | 3 days
  The occurence of postoperative cardiac arrhythmia the first three days following surgery, with cardiac arrhythmia defined as:
  * Atrial fibrillation (AF) or
  * Atrial Flutter (AFL) or
  * Ventricular Tachycardia (VT- both monomorphic and polymorphic types) or
  * Recurrent sustained ventricular tachycardia (RSVT) or
  * Ventricular fibrillation (VF) or
  * Torsade de Pointes (TDP) or
  * 2nd degree atrioventricular (AV) block or
  * 3rd degree atrioventricular (AV) block
The occurence of per- and postoperative ischemic ECG changes (until POD3) | 3 days
  The occurence of per- and postoperative ischemic ECG changes the first three days following surgery, defined as:
  * ST-depression ≥ 0,5 mm at the J-point in ≥ 2 contiguous leads or
  * Inverted T waves ≥ 1 mm in ≥2 contiguous leads that have dominant R waves or
  * ST-elevation ≥ 1 mm in ≥ 2 contiguous leads, however
  * ST-elevation in V2-V3 ≥ 2,5 mm for males < 40 years of age in ≥ 2 contiguous leads
  * ST-elevation in V2-V3 ≥ 2,0 mm for males ≥ 40 years of age in ≥ 2 contiguous leads
  * ST-elevation in V2-V3 ≥ 1,5 mm for females in ≥ 2 contiguous leads) or
  * In V2-V3: Any q wave ≥ 0,02 seconds,
  * In other leads: Q wave ≥ 0,03 seconds and > 1 mm deep in ≥ 2 contiguous leads.
The occurence of postoperative hypoxemia during the first three postoperative days | 3 days
  The occurence of postoperative hypoxemia during the first three postoperative days, defined as:
  * the number of declines in saturation of 4 % (or more) lasting 20 seconds (or more) or
  * number of desaturation episodes below 90 % or
  * time (minutes( spent below 90 %,

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Gögenur, MD, Study Chair — Zealand University Hospital; Jakob Burcharth, MD, Principal Investigator — Zealand University Hospital
Locations (1):
- Department of Surgery, Zealand University Hospital, Denmark., Køge, Denmark